CLINICAL TRIAL: NCT00047515
Title: Phase III Safety and Efficacy Study to Evaluate Combination IOP Lowering Therapy in Open Angle Glaucoma and Ocular Hypertensive Patients C-01-69.
Brief Title: Phase 3 Study to Evaluate IOP Lowering Therapy in Open Angle Glaucoma and Ocular Hypertension C-01-69
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-69; C-01-69
Record Dates: First submitted 2002-10-08; First posted 2002-10-18 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: open-angle; glaucoma; ocular; hypertension; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma; Hypertension

INTERVENTIONS:
Drug: Alcon Investigational Agent

SUMMARY:
To compare intraocular pressure lowering effectiveness of a combination drug vs. two individual drugs dosed alone.

ELIGIBILITY:
Adult subjects of either sex and any race with open-angle glaucoma or ocular hypertension; visual acuity of 20/80 to 20/400 or better (Snellen equivalent) or logMAR visual acuity not worse than 0.6. Clinically relevant ophthalmic or systemic conditions may be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Sites, Multiple Locations Throughout the United States, Texas, United States